CLINICAL TRIAL: NCT03472586
Title: Ipilimumab and Nivolumab in Combination With Immunoembolization for the Treatment of Metastatic Uveal Melanoma
Brief Title: Ipilimumab and Nivolumab With Immunoembolization in Treating Participants With Metastatic Uveal Melanoma in the Liver
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18P.042; JT 10364 (Other: JeffTrial Number)
Record Dates: First submitted 2018-03-14; First posted 2018-03-21 (Actual); Results first posted 2023-11-29 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Malignant Neoplasm in the Liver; Metastatic Uveal Melanoma; Stage IV Uveal Melanoma AJCC v7
MeSH Terms: conditions — Uveal Melanoma | interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab; Embolization, Therapeutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ipilimumab, nivolumab, immunoembolization) (Experimental): Patients receive ipilimumab IV over 30 minutes and nivolumab IV over 30 minutes on day 1. Patients also undergo immunoembolization on day 2. Cycles repeat every 3 weeks for 12 weeks in the absence of disease progression or unacceptable toxicity. Patients with complete response, partial response, or stable disease may receive nivolumab IV on day 1 and undergo immunoembolization on day 2. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. The interval between treatments may be extended up to every 6 weeks at the discretion of the treating physician.
  Interventions: Biological: Ipilimumab; Biological: Nivolumab; Drug: Embolization Therapy

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; 720801; 477202-00-9; 732442
Biological: Nivolumab — Given IV
  Other Names: 946414-94-4; BMS-936558; ONO-4538; Opdivo
Drug: Embolization Therapy — Undergo immunoembolization

SUMMARY:
This phase II trial studies ipilimumab and nivolumab with immunoembolization in treating patients with uveal melanoma that has spread to the liver. Immunotherapy with monoclonal antibodies, such as ipilimumab and nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Immunoembolization may kill tumor cells due to loss of blood supply and develop an immune response against tumor cells. Giving ipilimumab and nivolumab with immunoembolization may work better in treating patients with uveal melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the clinical benefit of treatment with immunoembolization (IEMBO) in combination with ipilimumab and nivolumab.

SECONDARY OBJECTIVES:

I. Determine all treatment and immune related toxicities. II. Determine progression free survival. III. Determine overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic uveal melanoma in the liver; patients must have at least one measurable liver metastasis that is >= 10 mm in longest diameter by computed tomography (CT) scan or magnetic resonance imaging (MRI)
* The total volume of the tumors must be less than 50% of the liver volume
* Willingness and ability to give informed consent
* Agreement to access archival tissue or agreement for tumor biopsy prior to treatment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, or 1
* Serum creatinine =< 2.0 mg/dl
* Granulocyte count >= 1000/mm^3
* Platelet count >= 100,000/mm^3
* Bilirubin =< 2.0 mg/ml
* Albumin >= 3.0 g/dl
* Prothrombin time (PT)/partial thromboplastin time (PTT) less than 1.5 times normal
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 3 x upper limit of normal (ULN)
* Alkaline phosphatase less than 1.5 times ULN (grade 1)
* Women must not be pregnant or breast-feeding
* Women of child-bearing potential must use at least two other accepted and effective methods of contraception and/or to abstain from sexual intercourse for at least 23 weeks after the last dose of nivolumab and/or ipilimumab and sexually active males must use at least two other accepted and effective methods of contraception and/or to abstain from sexual intercourse for at least 31 weeks after the last dose of nivolumab and/or ipilimumab

Exclusion Criteria:

* Failure to meet any of the criteria set forth in the inclusion criteria section
* Previous systemic exposure to anti-CTLA-4 antibody or anti-PD1 antibody
* Previous liver-directed treatments including chemoembolization, radiosphere, hepatic arterial perfusion, or drug-eluting beads; liver resection and focal ablation are permitted
* Presence of symptomatic liver failure including ascites and hepatic encephalopathy
* Presence of untreated brain metastases; if patients have had previous treatment for the brain metastasis, an MRI or CT scan of the brain must confirm the stabilization of the brain metastasis for more than 2 months
* Presence of uncontrolled hypertension or congestive heart failure, or acute myocardial infarction within 6 months of entry
* Presence of any other medical complication that implies survival of less than six months
* Uncontrolled severe bleeding tendency or active gastrointestinal (GI) bleeding
* Significant allergic reaction to contrast dye or granulocyte-macrophage colony-stimulating (GM-CSF)
* Immunosuppressive treatments within 4 weeks prior to embolization, unless prednisone =< 5 mg or equivalent
* Pregnancy or breast-feeding women
* Patients with active hepatitis with serum glutamic-oxaloacetic transaminase (SGOT) and serum glutamate pyruvate transaminase (SGPT) equal or greater than 5 times normal
* Biliary obstruction, biliary stent or prior biliary surgery except cholecystectomy
* Positive for known human immunodeficiency virus (HIV) Infection
* Uncontrolled chronic obstructive pulmonary disease or previous known pulmonary fibrosis
* Active infection
* Auto-immune disease including inflammatory bowel disease, lupus, rheumatoid arthritis, but not including hypothyroidism or psoriasis if condition has been stable for 2 months or greater

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marlana Orloff, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Sidney Kimmel Cancer Center at Thomas Jefferson University — https://www.jeffersonhealth.org/clinical-specialties/cancer
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Ipilimumab, Nivolumab, Immunoembolization)
Started | 14
Completed | 1
Not Completed | 13
Not completed — Physician Decision | 6
Not completed — Death | 6
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ipilimumab, Nivolumab, Immunoembolization)
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Hepatic Metastasis Stabilization Rate by Response Criteria (Response Evaluation Criteria in Solid Tumors [RECIST] 1.1)
Description: Defined as complete response + partial response + stable disease. Rated by Response Evaluation Criteria in Solid Tumors version 1.1. The estimate of the hepatic metastasis stabilization rate will be presented with corresponding 95% confidence intervals. The method of Atkinson and Brown will be used to adjust for the two-stage design.
Time Frame: At the end of 4th treatment cycle (Day 84 +/- 3 days). Cycles are 21 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ipilimumab, Nivolumab, Immunoembolization)
Number analyzed (Participants) | 14
Participants
  Complete response | 0
  Partial response | 0
  Stable Disease | 8
  Progressive disease | 5
  Not Evaluated | 1

2. Secondary Outcome: Incidence of Adverse Events
Description: Graded by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. Toxicity rates will be estimated with corresponding 95% confidence intervals.
Time Frame: Up to 1 year
Reporting Status: Not Posted

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Will be estimated using the Kaplan-Meier method.
Time Frame: From the start of the treatment to confirmation of progression of disease, assessed up to 1 year
Reporting Status: Not Posted

4. Secondary Outcome: Overall Survival
Description: Will be estimated using the Kaplan-Meier method.
Time Frame: From the start of the treatment to confirmation of progression of disease, assessed up to 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The adverse event reporting period for this trial begins when the patient receives the first treatment and ends 3 months after completion or withdrawal from the study. Treatment period is maximum of 2 years, thus reporting period is maximum of 27 months.
Arm/Group | Treatment (Ipilimumab, Nivolumab, Immunoembolization)
All-Cause Mortality (participants affected / at risk) | 13/14
Serious Adverse Events (participants affected / at risk) | 1/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ipilimumab, Nivolumab, Immunoembolization) (N=14)
grade 3 thromboembolic event that resulted in a hospitalization (Vascular disorders) | 1 (1)
hepatic hemorrhage - grade 3 (Hepatobiliary disorders) | 1 (1)
Dyspnea - Grade 5 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Death (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Paresthesia - Grade 1 (Vascular disorders) | 1 (1)
Diarrhea - grade 3 (Gastrointestinal disorders) | 1 (1)
Colitis - grade 3 (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ipilimumab, Nivolumab, Immunoembolization) (N=14)
death - disease progression (General disorders) | 6 (6)
Tachycardia - Grade 1 (Cardiac disorders) | 1 (1)
Vertigo - Grade 0 (Ear and labyrinth disorders) | 13 (13)
Chills - 0 (General disorders) | 10 (10)
Fatigue - Grade 0 (Gastrointestinal disorders) | 7 (7)
Edema - extremities - grade 0 (General disorders) | 12 (12)
Pericardial Effusion - Grade 0 (Cardiac disorders) | 14 (14)
Tachycardia - Grade 0 (Cardiac disorders) | 13 (13)
Vertigo - Grade 1 (Ear and labyrinth disorders) | 1 (1)
Hyperthyroidism - Grade 0 (Endocrine disorders) | 14 (14)
Hypothyroidism - Grade 0 (Endocrine disorders) | 14 (14)
Blurred vision - Grade 0 (Eye disorders) | 14 (14)
Decreased vision - grade 0 (Eye disorders) | 14 (14)
Chills - Grade 1 (General disorders) | 2 (2)
Chills - Grade 2 (General disorders) | 2 (2)
Fatigue - Grade 1 (General disorders) | 4 (4)
Fatigue - Grade 2 (General disorders) | 3 (3)
Edema - extremities - Grade 1 (General disorders) | 2 (2)
Fever - Grade 0 (General disorders) | 7 (7)
Fever - Grade 1 (General disorders) | 5 (5)
Fever - Grade 2 (General disorders) | 2 (2)
Flu-like symptoms - Grade 0 (General disorders) | 12 (12)
Flu-like symptoms - Grade 1 (General disorders) | 2 (2)
Edema - Localized - Grade 0 (General disorders) | 12 (12)
Edema - Localized - Grade 1 (General disorders) | 2 (2)
Non-cardiac chest pain - Grade 0 (General disorders) | 10 (10)
Non-cardiac chest pain - Grade 1 (General disorders) | 4 (4)
Pain - Grade 0 (General disorders) | 11 (11)
Pain - Grade 1 (General disorders) | 1 (1)
Pain - Grade 2 (General disorders) | 1 (1)
Pain - Grade 3 (General disorders) | 1 (1)
Rigors - Grade 0 (General disorders) | 12 (12)
Rigors - Grade 1 (General disorders) | 1 (1)
Abdominal bloating - Grade 0 (Gastrointestinal disorders) | 14 (14)
Abdominal distension - Grade 0 (Gastrointestinal disorders) | 14 (14)
Abdominal pain - grade 0 (Gastrointestinal disorders) | 3 (3)
Abdominal pain - Grade 1 (Gastrointestinal disorders) | 9 (9)
Abdominal pain - Grade 2 (Gastrointestinal disorders) | 1 (1)
Abdominal pain - Grade 3 (Gastrointestinal disorders) | 1 (1)
Colitis - Grade 0 (Gastrointestinal disorders) | 14 (14)
Constipation - Grade 0 (Gastrointestinal disorders) | 14 (14)
Diarrhea - Grade 0 (Gastrointestinal disorders) | 14 (14)
Dry Mouth - Grade 0 (Gastrointestinal disorders) | 14 (14)
Dyspepsia - Grade 0 (Gastrointestinal disorders) | 13 (13)
Dysphagia - Grade 0 (Gastrointestinal disorders) | 14 (14)
Dyspepsia - Grade 1 (Gastrointestinal disorders) | 1 (1)
Flatulence - Grade 0 (Gastrointestinal disorders) | 14 (14)
Nausea - Grade 0 (Gastrointestinal disorders) | 5 (5)
Nausea - Grade 1 (Gastrointestinal disorders) | 6 (6)
Nausea - Grade 2 (Gastrointestinal disorders) | 3 (3)
Vomiting - Grade 0 (Gastrointestinal disorders) | 7 (7)
Vomiting - Grade 1 (Gastrointestinal disorders) | 2 (2)
Vomiting - Grade 2 (Gastrointestinal disorders) | 5 (5)
Hepatic Pain - Grade 0 (Hepatobiliary disorders) | 12 (12)
Hepatic Pain - Grade 2 (Hepatobiliary disorders) | 2 (2)
ALT increased - Grade 0 (Investigations) | 10 (10)
ALT increased - Grade 3 (Investigations) | 3 (3)
ALT increased - Grade 4 (Investigations) | 1 (1)
AST increased - Grade 0 (Investigations) | 10 (10)
AST increased - Grade 3 (Investigations) | 3 (3)
AST increased - Grade 4 (Investigations) | 1 (1)
Blood bilirubin increased - Grade 0 (Investigations) | 13 (13)
Blood bilirubin increased - Grade 3 (Investigations) | 1 (1)
Creatinine increased - Grade 0 (Investigations) | 13 (13)
Creatinine increased - Grade 1 (Investigations) | 1 (1)
Creatinine Kinase increased - Grade 0 (Investigations) | 14 (14)
Troponin Increased - Grade 0 (Investigations) | 14 (14)
Arthralgia - Grade 0 (Musculoskeletal and connective tissue disorders) | 14 (14)
Back pain - grade 0 (Musculoskeletal and connective tissue disorders) | 9 (9)
Back pain - Grade 1 (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain - Grade 2 (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain - Grade 3 (Musculoskeletal and connective tissue disorders) | 1 (1)
Gait disturbance - Grade 0 (Musculoskeletal and connective tissue disorders) | 13 (13)
Gait disturbance - Grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized Muscle Weakness - Grade 0 (Musculoskeletal and connective tissue disorders) | 14 (14)
Hand pain - Grade 0 (Musculoskeletal and connective tissue disorders) | 13 (13)
Hand pain - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Hip Pain - Grade 0 (Musculoskeletal and connective tissue disorders) | 13 (13)
Hip Pain - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee pain - Grade 0 (Musculoskeletal and connective tissue disorders) | 14 (14)
Muscle cramps - Grade 0 (Musculoskeletal and connective tissue disorders) | 13 (13)
Muscle cramps - Grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia - Grade 0 (Musculoskeletal and connective tissue disorders) | 14 (14)
Neck pain - Grade 0 (Musculoskeletal and connective tissue disorders) | 14 (14)
Shoulder pain - Grade 0 (Musculoskeletal and connective tissue disorders) | 12 (12)
Shoulder pain - Grade 1 (Musculoskeletal and connective tissue disorders) | 2 (2)
Anorexia - Grade 0 (Metabolism and nutrition disorders) | 12 (12)
Anorexia - Grade 2 (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia - Grade 0 (Metabolism and nutrition disorders) | 14 (14)
Hypoalbuminia - Grade 0 (Metabolism and nutrition disorders) | 14 (14)
Hyponatremia - Grade 0 (Metabolism and nutrition disorders) | 14 (14)
Hypophosphatemia - Grade 0 (Metabolism and nutrition disorders) | 13 (13)
Hypophosphatemia - Grade 3 (Metabolism and nutrition disorders) | 1 (1)
Weight loss - Grade 0 (Metabolism and nutrition disorders) | 13 (13)
Weight loss - Grade 1 (Metabolism and nutrition disorders) | 1 (1)
Dizziness - Grade 0 (Nervous system disorders) | 14 (14)
Dysgeusia - Grade 0 (Nervous system disorders) | 12 (12)
Dysgeusia - Grade 2 (Nervous system disorders) | 2 (2)
Headache - Grade 0 (Nervous system disorders) | 14 (14)
Larynsophageal Dysthesia - Grade 0 (Nervous system disorders) | 14 (14)
Paresthesia - Grade 0 (Nervous system disorders) | 13 (13)
Paresthesia - Grade 3 (Nervous system disorders) | 1 (1)
Peripheral Neuropathy - Grade 0 (Nervous system disorders) | 14 (14)
Postoperative hemorrhage - Grade 0 (Surgical and medical procedures) | 11 (11)
Postoperative hemorrhage - Grade 1 (Surgical and medical procedures) | 2 (2)
Postoperative hemorrhage - Grade 2 (Surgical and medical procedures) | 1 (1)
Confusion - Grade 0 (Psychiatric disorders) | 14 (14)
Scrotal edema - Grade 0 (Reproductive system and breast disorders) | 14 (14)
Urinary incontinence - Grade 0 (Renal and urinary disorders) | 14 (14)
Cough - Grade 0 (Respiratory, thoracic and mediastinal disorders) | 14 (14)
Dyspnea - Grade 0 (Respiratory, thoracic and mediastinal disorders) | 14 (14)
Pleural Effusion - Grade 0 (Respiratory, thoracic and mediastinal disorders) | 14 (14)
Erythematous Papule - Grade 0 (Skin and subcutaneous tissue disorders) | 14 (14)
Pain at cath. site - Grade 0 (Skin and subcutaneous tissue disorders) | 12 (12)
Pain at cath. site - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Pain at cath. site - Grade 2 (Skin and subcutaneous tissue disorders) | 1 (1)
Periorbital Edema - Grade 0 (Skin and subcutaneous tissue disorders) | 13 (13)
Periorbital Edema - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus - Grade 0 (Skin and subcutaneous tissue disorders) | 14 (14)
Rash - Maculopapular - Grade 0 (Skin and subcutaneous tissue disorders) | 14 (14)
Rash - Pustular - Grade 0 (Skin and subcutaneous tissue disorders) | 14 (14)
Skin Ulceration - Grade 0 (Skin and subcutaneous tissue disorders) | 14 (14)
Uticaria - Grade 0 (Skin and subcutaneous tissue disorders) | 14 (14)
Hematoma - Grade 0 (Vascular disorders) | 13 (13)
Hematoma - Grade 1 (Vascular disorders) | 1 (1)
Hypotension - Grade 0 (Vascular disorders) | 12 (12)
Hypotension - Grade 1 (Vascular disorders) | 1 (1)
Hypotension - Grade 2 (Vascular disorders) | 1 (1)
Thromboembolic event - Grade 0 (Vascular disorders) | 13 (13)
Thromboembolic event - Grade 3 (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT03472586/Prot_SAP_000.pdf